CLINICAL TRIAL: NCT04566315
Title: SYMPTOMATIC EFFECTIVENESS OF MICROPARTICLE ARTERIAL EMBOLIZATION IN PATIENTS WITH TOTAL KNEE PROSTHESIS WITH PAIN RESISTANT TO MEDICAL TREATMENT
Brief Title: EMBOLIZATION IN PATIENTS WITH TOTAL KNEE PROSTHESIS WITH PAIN RESISTANT TO MEDICAL TREATMENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-AOIP-04; 2020-A01447-32 (Other: ID RCB)
Record Dates: First submitted 2020-07-24; First posted 2020-09-28 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARTERIAL EMBOLIZATION IN PATIENTS WITH TOTAL KNEE PROSTHESIS (Other): SYMPTOMATIC EFFECTIVENESS OF MICROPARTICLE ARTERIAL EMBOLIZATION IN PATIENTS WITH TOTAL KNEE PROSTHESIS WITH PAIN RESISTANT TO MEDICAL TREATMENT
  Interventions: Procedure: Arteriography knee arteriography

INTERVENTIONS:
Procedure: Arteriography knee arteriography — arteriography and an injection of inert microparticles of 75 μm in neovessels

SUMMARY:
The objective of this study is to evaluate at 3 months in a prospective study, the effectiveness of arterial embolization of neo-vessels in patients with a painful total knee prosthesis despite a well-conducted medical treatment

DETAILED DESCRIPTION:
To date, no study has attempted to measure the effects of arterial embolization on pain in patients with total knee prosthesis. It would be interesting to evaluate, in a therapeutic trial with a good level of evidence, this alternative to drug treatments that are often poorly tolerated, contraindicated or failing in this population of elderly subjects often presenting co-morbidities. This pilot study will be used to calculate the number of patients to be included in a comparative, placebo-controlled, double-blind study. In addition to the evaluation of the undesirable effects of arterial embolization, the objective of this study is to evaluate the effectiveness at 3 and 6 months of embolization of the neovessels on pain, stiffness, physical activity, quality of life and consumption of analgesics and anti-inflammatories.

Evaluation criteria: modification of the pain item in the EVA (Analog Visual Scale), EQ-5D (quality of life scale), and Knee injury and Osteoarthritis Outcome Score (KOOS) self-questionnaire collected in the 15 days preceding the procedure and then at 3 and 6 months ; the use of analgesics and anti-inflammatories; adverse events.

Study population: Patients aged 40 to 80 years with a painful total knee joint. The visual analogue scale (VAS) score must be greater than or equal to 50 mm for at least 3 months optimal medical treatment, and for whom, no surgical retreatment is indicated.

The expected benefits are the improvement of the treatment of patients in therapeutic impasse, wearing a total knee prosthesis whose pain is rebellious and disabling. More generally, the investigators expect an improvement in the quality of life of these patients currently without satisfactory alternative care.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 40 to 80.
* Total knee joint or bilateral Pain with EVA ≥ 50 mm evolving for at least 3 months despite the initiation of a well conducted medical treatment according to current recommendations including analgesics, NSAIDs, rehabilitation and weight loss

Exclusion Criteria:

* Minor person.
* Protected adults under the law. Patients deprived of their liberties. Subject not cooperative or unable to meet the requirements of the protocol.
* Subject participating in another clinical trial or in period of exclusion from a previous clinical trial. Severe visceral failure.
* Local infection. Algoneurodystrophy.
* Prosthesis loosening.
* Pregnant or breastfeeding woman.
* Allergy to contrast media.
* Chronic or acute renal failure (clearance <30 ml / min).
* Hemostasis disorders (blood platelet count <50,000 / mm3 or patient TCA / control TCA> 1.2 or TP <50%).
* Operative indication for removal of the retained prosthesis.
* Patient with obliterating arterial disease of the lower limbs.
* Contraindication to lidocaine: Known hypersensitivity to lidocaine hydrochloride, to local amide anesthetics or to any of the excipients.
* Patients with recurrent porphyria

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Knee injury self-questionnaire | in the 15 days preceding the procedure
  modification of the pain item in the Knee injury self-questionnaire collected
Knee injury self-questionnaire | at 3 months
  modification of the pain item in the Knee injury self-questionnaire collected
Osteoarthritis Outcome Score (KOOS) self-questionnaire | in the 15 days preceding the procedure
  and Osteoarthritis Outcome Score (KOOS) self-questionnaire collected
Osteoarthritis Outcome Score (KOOS) self-questionnaire | at 3 months
  and Osteoarthritis Outcome Score (KOOS) self-questionnaire collected

SECONDARY OUTCOMES:
EVA (Analog Visual Scale) | in the 15 days preceding the procedure ,
  EVA (Analog Visual Scale) score from 0 to 10
EVA (Analog Visual Scale) | at 3 months
  EVA (Analog Visual Scale) score from 0 to 10
EVA (Analog Visual Scale) | at 6 months
  EVA (Analog Visual Scale) score from 0 to 10
Osteoarthritis Outcome Score (KOOS) self-questionnaire | in the 15 days preceding the procedure,
  KOOS
Osteoarthritis Outcome Score (KOOS) self-questionnaire | at 3 months,
  KOOS
Osteoarthritis Outcome Score (KOOS) self-questionnaire | at 6 months,
  KOOS
EQ-5D (quality of life scale) | in the 15 days preceding the procedure
  EQ-5D (quality of life scale)
EQ-5D (quality of life scale) | at 3 months,
  EQ-5D (quality of life scale)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Sedat, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, CHU de NICE, France

IPD SHARING:
Plan to Share IPD: No